CLINICAL TRIAL: NCT05903742
Title: Standardising Care for Hepatitis Delta in the Netherlands
Acronym: DREAM-2
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maag Lever Darm Stichting (Other)
Responsible Party: Principal Investigator, Milan Sonneveld, Principal investigator, Erasmus Medical Center
Other Study IDs: 10022
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis D
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatitis delta cohort: hepatitis delta patients aged ≥18 years

SUMMARY:
Rationale: Hepatitis delta virus (HDV) is a defective RNA virus that requires presence of hepatitis B virus (HBV) to complete virion assembly and secretion. HBV-HDV coinfection ("hepatitis delta") has been associated with severe liver injury that may result in rapid progression to cirrhosis and hepatic decompensation, as well as a higher risk of liver cancer when compared to patients with HBV mono-infection. Given the low incidence of hepatitis D, experience in caring for individuals with hepatitis delta is limited and management practices vary.

Objective: Generate prospective follow-up data to increase our understanding of this rare disease.

Study design: Prospective observational cohort study spanning 5 years, during which we will collect standard clinical data as well as blood samples and quality of life questionnaires.

Study population: hepatitis delta patients aged ≥18 years Intervention (if applicable): not applicable Main study parameters/endpoints: Incidence of liver related events (liver cancer, (decompensation of) cirrhosis, liver transplantation) during follow-up and changes in markers of viral replication, inflammatory activity and liver stiffness over time.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks associated with participation can be considered negligible and the burden can be considered minimal. The only additional action that the participants must perform are the filling out of two annual quality of life questionnaires, which are considered non-invasive, and collection of 10 ml blood during regular blood sample collections

ELIGIBILITY:
Inclusion Criteria:

* Active hepatitis delta based on a positive anti-HDV and a positive HDV-RNA test
* Patients must be ≥18 years
* Written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hepatitis delta patients currently in care at the participating sites will be asked to enter the study. The exact number of eligible patients is unclear, but based on the DREAM-1 study we expect to enrol up to 150 patients.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Prospective population based follow-up data | 5 year
  Generate prospective population based follow-up data of a homogeneously managed hepatitis delta cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No